CLINICAL TRIAL: NCT02456064
Title: Impact of a Program of Non-pharmacological Intervention in Patients With Type 2 Diabetes Mellitus With Poor Control of Their Disease
Brief Title: Impact of a Program of Non-pharmacological Intervention in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Equipo Multidisciplinar Sanitario CS Foietes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Equipo Multidisciplinar
Record Dates: First submitted 2015-05-24; First posted 2015-05-28 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle counseling (Experimental): In this group we will make an intensive program based on: workshops, educational talks, group medical practices and "expert patient" among others conduct auditions.
  Interventions: Behavioral: Lifestyle counseling
- Normal group (No Intervention): In this group will be controlled as usual in the consultations.

INTERVENTIONS:
Behavioral: Lifestyle counseling — * Group medical visits
  * Telephone medical consultations
  * Expert patient
  * Training workshops
  Arms: Lifestyle counseling

SUMMARY:
The purpose of this study is to determine whether a non-drug intensive program can help improve control of type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This study is based on the creation of two groups of patients with type 2 diabetes mellitus over a period of six months .

In one of the groups an intensive program be developed through : group medical consultations , workshops , informative talks, " expert patient " telephone inquiries .. etc. Meanwhile , the control group that will be followed in the consultations as usual.

We will make a determination of HbA1c at 3 months and 6 months later to assess whether there are significant differences between the two groups .

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus with poor control of their disease.
* No changes have been made in pharmacological previous 3 months.

Exclusion Criteria:

* Changes in their drug treatment in the past 3 months.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
HbA1c | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ivan S Silvera, Principal Investigator

IPD SHARING:
Plan to Share IPD: No